CLINICAL TRIAL: NCT00875810
Title: PRESTIGE Observational Study
Status: Completed | Type: Observational
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: PRESTIGE Observational Study
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Degenerative Cervical Disc Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prestige artificial disc replacement is an alternative treatment option with 16 years of experience addressing the unmet needs of surgical fusion interventions. Previous studies on the PRESTIGE® cervical disc have proven the safety and effectiveness of artificial disc surgery with level I evidence.

The PRESTIGE Observational Study is intended to collect prospectively observational data primarily on the Quality of Life (QoL).

DETAILED DESCRIPTION:
Degenerative cervical disc disease is associated with a very high burden to the patient and the society. If conservative treatment options fail, surgical interventions are the last treatment option.

Symptomatic disc degeneration leads to neck pain, which can radiate to the scapula and arm, with dumbness and tingling, and sometimes grasping and walking difficulties. At an advanced stage, muscle weakness can be observed in the nerve territory.

The quality of life and functionality of patients with therapy-resistant (conservatively treated) severe degeneration of the disc is greatly impaired, as they suffer from intense pain and thus disability. Patients of working age were significantly more impacted by their symptoms than older patients. They are no longer able to fully participate in everyday activities.

Cervical neck pain resulting from degenerative disc disease is associated with a major economic burden for payers.

Traditional cervical surgical decompressions and fusions are currently the most common treatment option. Despite good treatment success rates, fusions are associated with a negative impact on the normal kinematics of the spine, long recuperation times and long absence from work. Prestige artificial disc replacement is an alternative treatment option.

The PRESTIGE Observational Study is intended to collect information on Quality of Life (QoL) prior and after PRESTIGE® Cervical Disc surgery; data on pain prior of participation to the study, drug regiment and X-ray evaluation throughout the course of the study will be obtained. In addition adverse events and economic data will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be willing to sign a Patient Data Release Form.
* Patient with degenerative disc disease (DDD) who is scheduled to receive a PRESTIGE® Cervical Disc and fulfills the indications according to the product description.

Exclusion Criteria:

* Patient fulfills any contraindication according to the product description.
* Patient has not reached the age of legal consent according to local laws.
* Patient has diabetes.
* Patient has Body Mass Index (BMI) > 35.
* Patient has affected disc not between C3/C4 and C6/C7.
* Patient with instability of cervical spine.
* Patients who will receive extensive decompression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with degenerative disc disease (DDD) who are scheduled to receive a cervical arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2008-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Štulik, MUDr, Principal Investigator — University Clinic Motol
Locations (20):
- Czechia (2):
  - Hospital Plzen - Lochotin, Pilsen
  - University Clinic Motol, Prague
- Agia Olga Hospital, Athens, Greece
- National Center for Spinal Disorders, Budapest, Hungary
- Kuwait (2):
  - Al-Salam International Hospital, Kuwait City
  - Razi Hospital for Orthopedic Surgery, Kuwait City
- Poland (7):
  - Centrum Rehabilitacji im.prof.M.Weissa "STOCER", Konstancin-Jeziorna
  - Centrum Ksztalcenia I Rehabilitcji, Konstancin
  - Centrum Rehabilitacji im.prof. M.Weissa "STOCER", Konstancin
  - State Hospital- Wojewodzkie Centrum, Opole
  - Specialist Hospital Prof. Alfreda Sokolowskiego, Szczecin
  - Orthopaedic University Hospital in Zakopane, Zakopane
  - State Hospital- Szpital Wojewodzki, Zielona Góra
- King Faisal Specialist Hospital & Research Center, Jeddah, Saudi Arabia
- Serbia (5):
  - Neurosurgical Clinic KCS, Belgrade
  - Clinical Center Nis Neurosurgical Clinic, Niš
  - Clinical Center Niš, Niš
  - Clinical Center of Vojvodina Neurosurgical Clinic, Novi Sad
  - Clinical Center of Vojvodina, Novi Sad
- NsP Nové Zámky Hospital, Nové Zamky, Slovakia

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervical Arthroplasty + Prestige LP: All patients were subjected to a cervical spinal arthroplasty. A complete discectomy was performed and the PRESTIGE® LP Cervical Disc System was inserted to replace the damaged intervertebral disc.
Period: Overall Study
Arm/Group | Cervical Arthroplasty + Prestige LP
Started | 194
Implanted | 190
Discharged | 177
3 Months Follow up | 175
6 Months Follow up | 80
12 Months Follow up | 112
24 Months Follow up | 148
Completed | 148
Not Completed | 46
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 3
Not completed — Lost to Follow-up | 39
Not completed — Patient enroled but not implanted | 2
Not completed — Device explanted | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cervical Arthroplasty + Prestige LP
Number analyzed (Participants) | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 63
Region of Enrollment [Number; unit: participants]
  Serbia | 10
  Saudi Arabia | 11
  Hungary | 13
  Czech Republic | 44
  Slovakia | 28
  Poland | 83
  Kuwait | 1

OUTCOME MEASURES:

1. Primary Outcome: EQ-5D
Description: The primary objective is the documentation of QoL before and after cervical disc surgery using the PRESTIGE® Cervical Disc System. The QoL will be determined using the EQ-5D questionnaire and the Neck Disability Index (NDI).
  EQ-5D is an instrument for measuring health outcome and consists of five dimensions: mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression and a Visual Analog Scale that can be used as a quantitative measure of health as judged by the patient. Each dimension has 3 levels (no problems = 1, some problems = 2, and extreme problems = 3). The EQ-5D index has an upper limit of 1 that indicates full health (indicated by "no problem" in all domains), whereas 0 represents death. Scores worst than 0 are possible, implying that some health states may be worse than death.
Time Frame: 2 years
Population: As this is an observational study not all patients completed EQ-5D questionnaires, for this reason the number of participants analyzed is different from the number of patients in the Participant Flow.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cervical Arthroplasty + Prestige LP
Number analyzed (Participants) | 155
units on a scale
  Baseline | 0.59 (0.22)
  3 months Follow up | 0.78 (0.16)
  6 months Follow up | 0.77 (0.20)
  12 months Follow up | 0.80 (0.19)
  24 months Follow up | 0.76 (0.21)

2. Secondary Outcome: Duration of Pain Prior to Enrollment
Description: Documentation of duration of pain prior to enrollment
Time Frame: Baseline visit
Measure: Number; unit: percentage of patients with pain
Arm/Group | Cervical Arthroplasty + Prestige LP
Number analyzed (Participants) | 190
percentage of patients with pain
  patients with pain for 3-6 months before surgery | 22.1
  patients with pain for 6-12 months before surgery | 21.3
  patients with pain for >12 months before surgery | 37.4

3. Primary Outcome: Neck Disability Index (NDI) Score
Description: The primary objective is the documentation of QoL before and after cervical disc surgery using the PRESTIGE® Cervical Disc System. The QoL will be determined using the EQ-5D questionnaire and the Neck Disability Index (NDI).
  The NDI is a self-reported questionnaire designed to provide information on how neck pain affects the patient's ability to manage in everyday life. It contains questions on 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
  NDI results can be presented as a raw score or as a percent. When presenting it as a raw score, each section is scored on a 0 to 5 rating scale and the result is summarized to a total score with a maximum score of 50. This raw score can also be doubled and expressed as a percentage. Zero points or 0% means no activity limitations and 50 points or 100% means complete activity limitation.
Time Frame: 2 years
Population: As this is an observational study not all patients completed NDI questionnaires, for this reason the number of participants analyzed is different from the number of patients in the Participant Flow.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cervical Arthroplasty + Prestige LP
Number analyzed (Participants) | 155
units on a scale
  Baseline | 24.1 (8.6)
  3 months Follow up | 13.2 (8.9)
  6 months Follow up | 12.6 (10.2)
  12 months Follow up | 12.3 (10.0)
  24 months | 13.4 (10.3)

4. Secondary Outcome: Intervertebral Disc Space
Time Frame: 2 years
Population: As this is an observational study not all patients had images available for each visit, for this reason the number of participants analyzed is different from the number of patients in the Participant Flow.
Measure: Mean (Standard Deviation); unit: millimiters
Arm/Group | Cervical Arthroplasty + Prestige LP
Number analyzed (Participants) | 96
millimiters
  Baseline | 0.22 (0.07)
  3 months Follow up | 0.41 (0.15)
  6 months Follow up | 0.42 (0.16)
  12 months Follow up | 0.40 (0.14)
  24 months Follow up | 0.39 (0.13)

ADVERSE EVENTS:
Arm/Group | Cervical Arthroplasty + Prestige LP
Serious Adverse Events (participants affected / at risk) | 7/190
Other Adverse Events (participants affected / at risk) | 40/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervical Arthroplasty + Prestige LP (N=190)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 2 (3)
syndroma carpi radialis (Nervous system disorders) | 1 (1)
Arm pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Quervain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Thoracic spine discopathy (Nervous system disorders) | 1 (1)
Wound hematoma (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervical Arthroplasty + Prestige LP (N=190)
Neck, shoulder and arm pain (General disorders) | 24 (25)
Lumbar pain (General disorders) | 16 (18)

LIMITATIONS AND CAVEATS:
Low patient compliance at the 6 and 12 months follow up visits

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release. The sponsor will limit its review to the determination of whether Confidential Information is disclosed and to check for technical correctness.